CLINICAL TRIAL: NCT03226626
Title: Tumescent Anesthesia Antibiotic Delivery (TAAD) and SubQKath for Prevention of Surgical Site Infection, Thrombosis and Sepsis
Brief Title: Tumescent Anesthesia Antibiotic Delivery (TAAD)
Acronym: TAAD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HK Surgical, Inc. (Industry)
Collaborators: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TAAD
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Surgical Site Infection; Thrombosis; Sepsis
Keywords: Tumescent; Lidocaine; Epinephrine; Cefazolin; Metronidazole; Surgical Site Infection; Thrombosis; Sepsis; Prevention; Prophylaxis
MeSH Terms: conditions — Surgical Wound Infection; Thrombosis; Sepsis | interventions — 1,3,4,6-tetra-O-acetyl-2-azido-2-deoxyglucopyranose

STUDY DESIGN:
Intervention Model Description: Prospective Meta-Analysis Multicenter Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Persons making decision to categorize the outcome as either "Infection Occurred" or "No Infection Occurred" will be masked with respect to whether or not the subject received Standard pre-operative IV antibiotics alone or received both IV antibiotics and tumescent anesthesia & antibiotic delivery (TAAD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- IVAD (Active Comparator): IV antibiotic delivery (IVAD) alone as surgical site infection prevention. The intervention is IV antibiotics alone.
  Interventions: Drug: Tumescent Anesthesia and antibiotic delivery (TAAD) plus IVAD
- TAAD + IVAD (Experimental): Both subcutaneous tumescent anesthesia & antibiotic delivery (TAAD) and IVADThe The intervention is subcutanious and IV antibiotics
  Interventions: Drug: Tumescent Anesthesia and antibiotic delivery (TAAD) plus IVAD; Device: SubQKath

INTERVENTIONS:
Drug: Tumescent Anesthesia and antibiotic delivery (TAAD) plus IVAD — Concomitant tumescent anesthesia antibiotic delivery (TAAD) & Intravenous antibiotic delivery (IVAD).
  Other Names: SubQKath
Device: SubQKath — The device intervention consists of using the SubQKath device to provide subcutaneous delivery of antibiotics.
  Arms: TAAD + IVAD

SUMMARY:
This is a multicenter randomized clinical trial (RCT) comparing two modes of antibiotic delivery:

Control: Intravenous Antibiotic Delivery (IVAD) Treatment: IVAD + TAAD The Food & Drug Administration (FDA) has approved our Investigational New Drug (IND) application to conduct this RCT. An IND application was necessary because subcutaneous injection of antibiotics in general, and cefazolin and metronidazole in particular are considered to be "off-label". In addition, the tumescent formulation of cefazolin (1gm) and metronidazole (500mg/100ml) in a dilute solution of lidocaine (1gm), epinephrine (1mg) in 100ml and sodium bicarbonate (10mEq/10ml) added a 1000ml bag of 0.9% sodium chloride (total volume 1210ml) is also considered "off-label." This trial will also prospectively study the HK Surgical SubQKath, an over-the-needle subcutaneous catheter specifically designed to deliver relatively large volumes of a relatively dilute TAAD solution. The TAAD trial will document the safety and efficacy of the HK SubQKath

DETAILED DESCRIPTION:
Based on the approval of an investigational new drug (IND) application, the present clinical trial of TAAD of cefazolin and metronidazole has been approved by the Division of Anti-Infective Products (DAIP).

Despite the use of multiple interventions, surgical site infection (SSI) continues to be a significant problem. There is a need for an effective, accessible, inexpensive, simple, safe technique that reduces the risk of SSI. Intravenous antibiotic delivery (IVAD) using an over-the-needle intravenous (IV) catheter is the current standard mode of antibiotic delivery for SSI prevention.

1. Subcutaneous delivery of an antibiotics such as cefazolin and metronidazole is considered by the FDA to be off-label.
2. Subcutaneous infiltration of dilute a tumescent lidocaine solution (with or without antibiotics) at lidocaine dosages between 7mg/kg and 28mg/kg is off-label.
3. Subcutaneous infiltration of dilute antibiotic(s) in a tumescent lidocaine solution using a novel over-the-needle subcutaneous catheter (SubQKath), having holes distributed along most of the length of the cannula length, requires FDA 510(k) approval.

This multicenter randomized clinical trial (RCT) protocol is designed to

1. compare two modes of antibiotic delivery,
2. validate the safety of tumescent lidocaine at dosages up to 28mg/kg,
3. validate the safety of the SubQKath for tumescent anesthetic antibiotic delivery (TAAD).
4. This protocol is not a clinical trial comparing the effects of different drugs.
5. This RCT compares IVAD alone versus concomitant TAAD and IVAD (TAAD+IVAD).

TAAD using a novel over-the-needle subcutaneous catheter (SubQKath) by direct subcutaneous infiltration of dilute antibiotic(s) in a tumescent lidocaine & epinephrine solution is a novel mode of antibiotic delivery.

From a statistical perspective, this protocol describes an open label randomized clinical trial (RCT) with prospective multicenter meta-analytic statistical design using sequential data analysis with one stopping point.

We hypothesize that, compared to IVAD alone, TAAD+IVAD will be superior in terms of reducing the risk of SSI, as well as venous thromboembolism (VTE) and systemic inflammatory response syndrome (SIRS).

These three hypotheses are supported by two recently published free open access online journal articles describing the pharmacokinetics of tumescent lidocaine anesthesia (TLA) and the tumescent anesthesia antibiotic delivery (TAAD):

Klein JA, Jeske DR. Estimated Maximal Safe Dosages of Tumescent Lidocaine. Anesth Analg. 2016;122:1350-9.

Klein JA, Langman LJ. Prevention of Surgical Site Infections and Biofilms: Pharmacokinetics of Subcutaneous Cefazolin and Metronidazole in a Tumescent Lidocaine Solution. Plast Reconstr Surg Glob Open 2017; e1351.

TAAD provides subcutaneous interstitial antibiotic concentrations that are 10 to 100 times greater than the concentration that can be achieved by IV antibiotic delivery. The lidocaine serum concentration-time profile following TLA closely resembles a constant IV infusion of lidocaine. In animal studies IV lidocaine infusions decrease the incidence and severity of sepsis. TLA lidocaine also inhibits in-vivo platelet function while promoting excellent surgical hemostasis. (unpublished data, manuscript in progress).

The statistical design of this multicenter randomized clinical trial is robust and relies on prospective meta-analysis. Individual research sites will choose the targeted category of research subjects based on each site's population of surgical patients and the clinical interests and expertise of the participating surgeons.

Some research site may be sophisticated high-tech medical centers caring for the most difficult colorectal surgical patients at exceptionally high risk for SSI. Some research sites may be located in medically impoverished countries with limited surgical resources and very high rates of SSI. Other research sites may be focused on the care of patients in burn centers, trauma patients with contaminated wounds, military combat casualties with grossly contaminated wounds, or patients with infected median sternotomy wounds undergoing muscle flap repair.

Within any given research site all research subjects will be randomly assigned prospectively to have similar surgical procedures. However, the type of surgical procedure can vary from one research site to another.

Tumescent infiltration (TI) drug delivery involves subcutaneous infiltration relatively large volumes (1 to 2 liters or more) of a relatively dilute solution of epinephrine (≤1mg) in a liter of either 0.9% physiologic saline or a similar balanced salt solution such as lactated Ringer's solution. From a pharmacokinetic perspective, a dilute tumescent infiltration (TI) solution functions as a drug delivery vehicle. Tumescent infiltration (TI) drug delivery is a mode of drug delivery that has a pharmacokinetic profile distinct from intravenous (IV), intramuscular (IM), oral (PO) or transcutaneous delivery.

When a TI Solution is used as a vehicle to deliver lidocaine subcutaneously we have TI solution + Lidocaine = tumescent lidocaine anesthesia (TLA). Further, when an antibiotic is added to a TLA solution, TI Solution + Lidocaine + Antibiotic, the result is a tumescent anesthetic antibiotic delivery (TAAD) solution.

Tumescent subcutaneous drug delivery provides

1. High and prolonged (12 to 18 hours or more) localized subcutaneous drug concentrations,
2. Slow steady systemic (serum) drug delivery having a concentration-time profile similar to a slow constant IV infusion and
3. A peak serum drug concentration that is substantially less than would be expected by routine doses given by IV delivery.
4. The antibiotic dilution and lidocaine of a TAAD solution avert both the potential tissue toxicity and pain associated direct subcutaneous injections of antibiotic at concentrations of commercial formulations intended for IV delivery.

TAAD can achieve subcutaneous antibiotic concentrations that exceed by more than 10-fold the subcutaneous concentrations achievable by IVAD. TAAD has the potential to prevent or overcome an antibiotic-resistant infection of subcutaneous tissue using less than the usual total mg IV dose of an antibiotic while providing higher subcutaneous antibiotic concentrations than can be achieved by IV delivery, and simultaneously avoid systemic antibiotic toxicity by limiting the rate of systemic antibiotic absorption and thus minimizing the peak antibiotic serum concentration.

For example, TAAD delivery of an aminoglycoside antibiotic has the potential to provide subcutaneous antibiotic concentrations that are sufficiently diluted to avoid local tissue toxicity while simultaneously providing subcutaneous antibiotic concentrations that are significantly higher than can be achieved by IV delivery, with a reduced risk of systemic (ear or kidney) toxicity.

The present research protocol, only allows the use of antibiotics that have FDA approval. Cefazolin and metronidazole have FDA approval for IV delivery. Both cefazolin and metronidazole are known to be safe and effective when delivered by subcutaneous infiltration as documented by published reports in peer-reviewed literature.

For antibiotics, the therapeutic benefits of IV delivery are muted by the fact that IV delivery often results in sub-therapeutic subcutaneous antibiotic concentrations and the associated increased risk of developing drug resistance. For some cutaneous infections and for preventing surgical site infections, tumescent infiltration drug delivery overcomes these limitations of IV delivery.

Scientific Generalizability This protocol is not a clinical trial comparing the effects of different drugs. This clinical trial protocol is designed to compare two modes of antibiotic delivery.

In order to maximize the generalizability of the results of this research, the protocol is designed to accommodate a wide variety of clinical situations encountered internationally. The protocol provides for the inclusion of a wide variety of pathology, surgical techniques, surgeon training/experience, quality of surgical facilities, diverse local health, local nutrition and local economic conditions. The protocol specifically allows for the use of locally available antibiotic products. Individual research sites will use their usual and customary sources of cefazolin, metronidazole, lidocaine, epinephrine, sodium bicarbonate and physiologic salt solutions.

Research sites will be provided with sufficient supply of devices (SubQKaths, tumescent lidocaine anesthesia (TLA) peristaltic pump and tubing) to facilitate efficient TAAD infiltration.

For the purposes of scientific validity and generalizability, this research intentionally does not restrict the choice of generic antibiotic to that of a single specified manufacturer. This protocol explicitly allows the use of any generic version of the antibiotic, irrespective of the manufacturer. This protocol also allows TAAD of an antibiotic that is only available as a branded (non-generic) drug.

In some cases, the principal investigator (PI) will supply individual research sites in medically indigent communities with a TAAD Drug Kit containing antibiotics, lidocaine with epinephrine, sodium bicarbonate and 1 liter bags of a balanced salt solution.

For the purpose of statistical analysis and validity, for any given subject, the same antibiotic(s) will be used for both TAAD and IVAD.

Within any individual research site, it is preferred that the antibiotic formulation, source and brand will be standardized and invariant, subject to continued availability of the antibiotic.

"Off-Label" Aspects of Tumescent Drug Delivery

The use of TAAD involves:

1. Subcutaneous antibiotic injection is "off-label" for most FDA-approved antibiotics.
2. The very dilute formulation of the antibiotic solution for TAAD is unapproved by the FDA.
3. The recommended maximum dosages for tumescent lidocaine (28mg/kg) is unapproved.

Primary and Secondary End Points This protocol is designed to prospectively collect data to evaluate the efficacy and safety of the TAAD mode of subcutaneous antibiotic delivery.

This protocol is designed to prospectively collect observational data to evaluate the safety and efficacy of the devices (HK SubQKath, HK tumescent infiltration tubing and HK peristaltic tumescent infiltration pumps) used for subcutaneous tumescent infiltration of TAAD solutions.

The primary end-point is the incidence of surgical site infections (SSI). The protocol compares TAAD + IVAD with IVAD alone with respect to:

1. the incidence of SSI,
2. the incidence of post-operative venous thromboembolism (VTE) and
3. the incidence of sepsis (pathogen-related or damage-related). The protocol also records device-related incidence of adverse events. The devices used for TAAD include a new single use subcutaneous infiltration cannula (HK SubQKath) for the tumescent drug delivery, tumescent peristaltic pumps and tumescent infiltration tubing.

Definitions: Tumescent anesthesia antibiotic delivery (TAAD) is defined as the subcutaneous infiltration of a dilute solution of antibiotic(s) in a solution of tumescent lidocaine anesthesia (TLA). TLA consists of a dilute solution of lidocaine (≤1gm/L), epinephrine (≤1mg/L) and sodium bicarbonate (10mEq/L) in 0.9% physiologic saline or lactated Ringer's solution. Our estimated maximal safe dosage of TLA lidocaine is 28mg/kg without liposuction.

We hypothesize that TAAD together with intravenous antibiotic delivery (IVAD) will significantly reduce the incidence of surgical site infections (SSI).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects greater than 18 years of age scheduled for surgical procedures considered to have a high risk for a surgical site infection (SSI) such as 1) secondary repair of a ventral hernia, 2) open bariatric surgery, 3) open abdominal colorectal surgery, 4) trauma surgery, 5) burn surgery or 6) sternotomy.
2. Patients ought to have one of the following risk factors for surgical site infection: emergency surgery, obesity, diabetes mellitus, cancer surgery, be immune-compromised or otherwise be at an increased risk for SSI, or be in a medically indigent environment where surgical aseptic technique is suboptimal

Exclusion Criteria:

Pre-existing skin infection Pregnant Less than 18 years old

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
surgical site infection (SSI) | within 30 of surgical procedure
  Occurrence of a surgical site infection (SSI)
Post-operative venous thromboembolism | within 30 of surgical procedure
  Diagnosis of Post-operative venous thromboembolism
Sepsis | within 30 of surgical procedure
  Diagnosis of Post-operative sepsis
Adverse event associated with SubQKath device | within 30 of surgical procedure
  any adverse event

SECONDARY OUTCOMES:
Length of Stay (LOS) in hospital after surgery (hours) | 60 days
  Length of Stay (LOS) in hospital after surgery (hours)
Time in post-operative/post-anesthesia recovery unit. | 30 days post-op
  Time in post-operative/post-anesthesia recovery unit.
Post-Op Narcotic Requirements (total mg and mg/kg) | 30 days post op
  Post-Op Narcotic Requirements (total mg and mg/kg) will be recorded.
General Anesthesia Requirements (Quantitative Measure) | day of surgery
  Quantitative measures of General Anesthesia Requirements (Quantitative Measure)
Diagnosis of C. Difficile colitis | 30 Days Postop
  Antibiotic related diarrhea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein JA, Jeske DR. Estimated Maximal Safe Dosages of Tumescent Lidocaine. Anesth Analg. 2016 May;122(5):1350-9. doi: 10.1213/ANE.0000000000001119. PMID 26895001
- [Background] Klein JA, Langman LJ. Prevention of Surgical Site Infections and Biofilms: Pharmacokinetics of Subcutaneous Cefazolin and Metronidazole in a Tumescent Lidocaine Solution. Plast Reconstr Surg Glob Open. 2017 May 30;5(5):e1351. doi: 10.1097/GOX.0000000000001351. eCollection 2017 May. PMID 28607871
- See also: Information about subcutaneous tumescent drug delivery — http://tumescent.org